CLINICAL TRIAL: NCT00639444
Title: Infant Nutrition and Development of Celiac Disease in Genetically At-risk Babies: a Dietary Intervention Study at Weaning
Brief Title: Risk of Celiac Disease and Age at Gluten Introduction
Acronym: CELIPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Associazione Italiana Celiachia (AIC) (Other); Menarini Group (Industry)
Responsible Party: Principal Investigator, Carlo Catassi, M.D., Associate Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPM-CE 204332
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten free diet (Active Comparator): the intervention in this group is keeping a gluten-free diet from 0 to 12 months
  Interventions: Dietary Supplement: gluten-free, normocaloric diet from 6 to 12 months
- Gluten containing diet (No Intervention): infants in this group are started on gluten-containing cereals at 6 months (control group)

INTERVENTIONS:
Dietary Supplement: gluten-free, normocaloric diet from 6 to 12 months — Gluten-containing cereals (wheat, rye and barley) will be replaced by gluten-free starchy food (rice, corn, tapioca-based, etc) in a normocaloric diet
  Other Names: gluten-free products
  Arms: Gluten free diet

SUMMARY:
The purpose of this study is to determine whether age at introduction of gluten-containing cereals (e.g. wheat) plays a role in influencing the risk of celiac disease (CD) development in infants with a first-degree relative affected by CD.

DETAILED DESCRIPTION:
We undertook a prospective study to establish the incidence of CD autoimmunity related to the timing of gluten exposure in at-risk infants. Infants at family risk for CD (at least one first-degree relative affected) are enrolled in this prospective, multicentre, intervention study conducted in Italy. Infants are randomly assigned to introduce gluten at either 4-6 or 12 months (groups A and B, respectively) and then enter a follow-up period of 5 years. Duration of breastfeeding and types of formulas, adherence to the dietary plan, amount of gluten administered, and clinical data are collected by phone or direct interview at 4, 7, 9, and 12 months of age. HLA (Human Leucocyte Antigene) status and CD serology (anti-transglutaminase and other autoantibodies) are tested at 15, 24, 36 and 60 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Newborn in a family where a first-degree relative is already affected with biopsy-proven CD

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 703 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
prevalence of active CD | 5 years of age

SECONDARY OUTCOMES:
prevalence of CD-related autoantibodies (IgA anti-transglutaminase) | age 2, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, MD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Department of Pediatrics, via Corridoni 11, Ancona, Italy

REFERENCES:
- [Background] Lionetti E, Castellaneta S, Pulvirenti A, Tonutti E, Francavilla R, Fasano A, Catassi C; Italian Working Group of Weaning and Celiac Disease Risk. Prevalence and natural history of potential celiac disease in at-family-risk infants prospectively investigated from birth. J Pediatr. 2012 Nov;161(5):908-14. doi: 10.1016/j.jpeds.2012.05.008. Epub 2012 Jun 15. PMID 22704250
- [Derived] Lionetti E, Castellaneta S, Francavilla R, Pulvirenti A, Tonutti E, Amarri S, Barbato M, Barbera C, Barera G, Bellantoni A, Castellano E, Guariso G, Limongelli MG, Pellegrino S, Polloni C, Ughi C, Zuin G, Fasano A, Catassi C; SIGENP (Italian Society of Pediatric Gastroenterology, Hepatology, and Nutrition) Working Group on Weaning and CD Risk. Introduction of gluten, HLA status, and the risk of celiac disease in children. N Engl J Med. 2014 Oct 2;371(14):1295-303. doi: 10.1056/NEJMoa1400697. PMID 25271602